CLINICAL TRIAL: NCT01219374
Title: A Longitudinal Prospective Study of Ovum Donors After Donation
Brief Title: Study of Ovum Donors After Donation
Status: Completed | Type: Observational
Sponsor: Reproductive Medicine Associates of New Jersey (Other)
Responsible Party: Sponsor
Other Study IDs: RMA-00-08
Record Dates: First submitted 2010-10-08; First posted 2010-10-13 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: Anonymous Donors
Keywords: egg donor

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- egg donors: anonymous egg donors

SUMMARY:
To explore the attitudes and reactions of ovum donors prospectively after ovum donation and to follow their medical histories.

DETAILED DESCRIPTION:
Although several studies have explored donor's reactions and experiences up to a year post donation, no study has explored how donor attitudes and reactions change over time. Currently, there is no long-term data available to describe donor's feelings and reactions to their donation. Consequently, programs have no guidance to counsel prospective donors about whether donors' attitudes change towards their own participation, contact with any offspring, or concerns about the donation. In addition, just as ovum donors' initial health histories were shared anonymously with the recipient(s), any updated information gathered in this study would be shared anonymously with the recipient(s) or offspring should they request those updates.

ELIGIBILITY:
All anonymous egg donors are eligible for participation.

Ages: 21 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Anonymous egg donors
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2006-12; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Do recipients' attitudes and reactions change over time regarding the selection criteria for their donors? | 12-15 Months
  Analysis of recipients' attitudes and reactions at initial psychoeducational consultation, a week after the initial psychoeducational consultion, at donor match and 3 months after delivery

CONTACTS AND LOCATIONS:
Overall Officials: Andrea M Braverman, PhD, Principal Investigator — Reproductive Medicine Associates of New Jersey
Locations (1):
- Reproductive Medicine Associates of New Jersey, Morristown, New Jersey, United States